CLINICAL TRIAL: NCT01153672
Title: A Pilot Study of Vorinostat to Restore Sensitivity to Aromatase Inhibitor Therapy
Brief Title: Vorinostat in Treating Patients With Stage IV Breast Cancer Receiving Aromatase Inhibitor Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hannah Linden, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6856; NCI-2010-01289 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-06-22; First posted 2010-06-30 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Vorinostat; Biopsy; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Anastrozole; Letrozole; exemestane; Gene Expression Profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (enzyme inhibitor therapy, AI sensitization therapy) (Experimental): Patients receive vorinostat PO QD for 2 weeks followed by AI therapy comprising anastrozole PO QD, letrozole PO QD, OR exemestane PO QD for 6 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Other: laboratory biomarker analysis; Procedure: biopsy; Radiation: F-18 16 alpha-fluoroestradiol; Procedure: positron emission tomography; Drug: anastrozole; Drug: letrozole; Drug: exemestane; Genetic: gene expression analysis

INTERVENTIONS:
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: laboratory biomarker analysis — Correlative studies
Procedure: biopsy — Optional correlative studies
  Other Names: biopsies
Radiation: F-18 16 alpha-fluoroestradiol — Correlative studies
  Other Names: F-18 FES; fluorine-18 16 alpha-fluoroestradiol
Procedure: positron emission tomography — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Drug: anastrozole — Given PO
  Other Names: ANAS; Arimidex; ICI-D1033
Drug: letrozole — Given PO
  Other Names: CGS 20267; Femara; LTZ
Drug: exemestane — Given PO
  Other Names: Aromasin; FCE-24304; PNU 155971
Genetic: gene expression analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies vorinostat in treating patients with stage IV breast cancer receiving aromatase inhibitor (AI) therapy. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Vorinostat may also help AI therapy work better by making tumor cells more sensitive to the drug

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the rate of clinical benefit (objective response plus stable disease) for patients treated with cycles consisting of 2 weeks of vorinostat followed by 6 weeks of AI therapy.

SECONDARY OBJECTIVES:

I. Assess the safety and tolerability of vorinostat in patients with metastatic breast cancer.

II. Assess the change in estrogen receptor (ER) expression, measured as the change in fluoroestradiol standard uptake value (FES SUV) using fluoroestradiol-positron emission tomography (FES-PET) completed per protocol 7184 after two weeks of vorinostat therapy and after 8 weeks of therapy.

III. Assess tumor metabolic response, measured as the change in fluorodeoxyglucose (FDG) SUV using FDG PET completed per protocol 7184 after two weeks of vorinostat therapy and after 8 weeks of therapy.

IV. Assess the change in hormone levels (estradiol, estrone, follicle-stimulating hormone [FSH], sex binding globulin, testosterone, and free testosterone) after 8 weeks of therapy.

V. Assess the change in ER, progesterone receptor (PR), human epidermal growth factor receptor 2 (HER2), androgen receptor (AR), epithelial growth factor receptor (EGFR), vascular endothelial growth factor (VEGF) tumor expression after two weeks of vorinostat therapy in patients that consent to optional tissue biopsy procedure.

VI. Assess the time to progression and the overall survival of patients treated with cycles of 2 weeks of vorinostat followed by 6 weeks of AI.

OUTLINE:

Patients receive vorinostat orally (PO) once daily (QD) for 2 weeks followed by AI therapy comprising anastrozole PO QD, letrozole PO QD, OR exemestane PO QD for 6 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months until disease progression, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of breast cancer
* Stage IV disease
* Patient has previously derived clinical benefit from endocrine therapy, but is no longer deriving benefit to endocrine therapy in the opinion of the treating investigator; patients need to stop AI for at least one week prior to starting vorinostat treatment on this protocol
* At least one site of measurable disease, as defined by the modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Female patient is post menopausal as defined by one of the following; free from menses for > 2 years, surgically sterilized ,FSH and Estradiol in post-menopausal range AND surgical absence of uterus OR chemotherapy induced amenorrhea lasting > 1 year OR currently on ovarian suppression
* Female patient of childbearing potential has a negative urine or serum (beta-human chorionic gonadotropin [hCG]) pregnancy test within 14 days prior to receiving the first dose of vorinostat
* Male patient agrees to use two barrier methods of contraception or abstain from intercourse for the duration of the study
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Prothrombin Time or international normalized ratio (INR) =< 1.5 x upper limit of normal (ULN) unless receiving therapeutic anticoagulation
* Partial thromboplastin time (PTT) =< 1.2 times the ULN unless the patient is receiving therapeutic anticoagulation
* Potassium and magnesium levels within normal limits
* Calculated creatinine clearance >= 30 mL/min
* Serum total bilirubin =< 1.5 X ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X ULN
* Alkaline Phosphatase =< 2.5 X ULN
* Patient, or the patient's legal representative, has voluntarily agreed to participate by giving written informed consent
* Patient has a life expectancy of at least 12 weeks in the opinion of the treating investigator
* Patient is willing to continue on same AI therapy
* Patient agrees to participate in imaging Protocol 7184 and is separately consented

Exclusion Criteria:

* Patient has not derived clinical benefit from prior endocrine therapy
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of initial dosing with study drug(s) other than the imaging protocol 7184
* Patient has received an ER blocking therapy (selective estrogen receptor modulating [SERM] or downregulating [SERD] i.e. tamoxifen or fulvestrant) within the past 6 weeks
* Patient had prior treatment with an histone deacetylase (HDAC) inhibitor (e.g., romidespin [Depsipeptide], NSC-630176, MS 275, LAQ-824, belinostat [PXD-101], LBH589, MGCD0103, CRA024781, etc); patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study; patients who have received such compounds for other indications, e.g. valproic acid for epilepsy, may enroll after a 30-day washout period
* Patient is on any systemic steroids that have not been stabilized to the equivalent of =<10 mg/day prednisone during the 30 days prior to the start of the study drugs
* Patient has known hypersensitivity to the components of study drug or its analogs
* Patients with uncontrolled brain metastases
* New York Heart Association (NYHA) Class III or IV congestive heart failure, myocardial infarction within the previous 6 months, corrected QT interval (QTc) > 0.47 seconds, or uncontrolled arrhythmia.
* Type I Diabetes Mellitus; patients with Type II Diabetes Mellitus will be included as long as their glucose can be controlled to under 200 mg/dL
* Patient is pregnant or breast feeding, or expecting to conceive or father children within the projected duration of the study
* Patient with a "currently active" second malignancy, other than non-melanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled; patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for > 5 years or are considered by their physician to be at less than 30% risk of relapse
* Patients with known active viral hepatitis
* Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study or is not in the best interest of the patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2016-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Linden, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy, AI Sensitization Therapy)
Started | 8
Completed | 6
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy, AI Sensitization Therapy)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Clinical Benefit According to RECIST
Description: Conventional imaging (CT, bone scan) was performed at baseline and at week 8 and tumor response assessed by RECIST criteria
Time Frame: Up to approximately 5 years
Measure: Number (90% Confidence Interval); unit: percentage of evaluable participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy, AI Sensitization Therapy)
Number analyzed (Participants) | 8
percentage of evaluable participants | 15 [12 to 65]

2. Primary Outcome: Duration of Response
Description: Duration of response will be summarized for responders.
Time Frame: Up to approximately 5 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Enzyme Inhibitor Therapy, AI Sensitization Therapy)
Number analyzed (Participants) | 2
weeks | 25.4 [18.3 to 32.4]

3. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier survival curves will be used to describe progression-free survival. For progression-free survival, patients without documented disease progression or death will be treated as censored observations on the date of the last tumor assessment.
Time Frame: Time elapsed from the first day of study treatment, until disease progression or death, assessed up to approximately 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy, AI Sensitization Therapy)
Number analyzed (Participants) | 8
months | 2.8 [1.9 to 13.3]

4. Secondary Outcome: Overall Survival
Description: Kaplan-Meier survival curves will be used to describe overall survival. Overall survival time will be censored on the last date the patient was known to be alive.
Time Frame: Time elapsed from the first day of study treatment until death, assessed up to approximately 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy, AI Sensitization Therapy)
Number analyzed (Participants) | 8
months | 28.8 [16.2 to 54.5]

5. Secondary Outcome: Percentage of Patients That Experience Adverse Events as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Time Frame: Up to approximately 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy, AI Sensitization Therapy)
Number analyzed (Participants) | 8
percentage of participants | 37.5

ADVERSE EVENTS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy, AI Sensitization Therapy)
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzyme Inhibitor Therapy, AI Sensitization Therapy) (N=8)
Flu-like symptoms (Infections and infestations) | 1 — Not related to study treatment
pancreatitis (Gastrointestinal disorders) | 1 — Not related to study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzyme Inhibitor Therapy, AI Sensitization Therapy) (N=8)
Fatigue (General disorders) | 2 — Grade 3 (CTCAE v3.0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes